CLINICAL TRIAL: NCT06181006
Title: A Phase I, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LOXO-305 in Healthy Adult Subjects
Brief Title: A Study to Evaluate Pirtobrutinib (LOXO-305) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20017; J2N-OX-JZNS (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: 300 mg Pirtobrutinib (Experimental): Participants received a single dose of Pirtobrutinib 300 milligram (mg) administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Cohort 2: 600 mg Pirtobrutinib (Experimental): Participants received a single dose of Pirtobrutinib 600 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Cohort 3: 800 mg Pirtobrutinib (Experimental): Participants received a single dose of Pirtobrutinib 800 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Cohort 4: 900 mg Pirtobrutinib (Experimental): Participants received a single dose of Pirtobrutinib 900 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of pirtobrutinib and to look at the amount of the study drug, pirtobrutinib, that gets into the blood stream and how long it takes the body to get rid of it when given in healthy adult participants. For each participant, the total duration of the study will be 46 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 8-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor

* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening or Check-in (Day -1)
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously completed or withdrawn from any other study investigating Pirtobrutinib (LOXO-305) and have previously received the investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Started | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Cohort 1: 300 mg Pirtobrutinib: Participants received a single dose of Pirtobrutinib 300 mg administered orally on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.79) | 36.2 (9.15) | 33.2 (10.85) | 35.3 (5.47) | 36.6 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 0 | 2 | 8
  Male | 2 | 4 | 6 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 3 | 15
  Not Hispanic or Latino | 2 | 0 | 4 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 2 | 7
  White | 4 | 5 | 3 | 3 | 15
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs)
Description: TEAE is defined as an adverse event (AE) which starts on or after the first administration of study drug. A serious adverse event is defined as any AE occurring at any dose that results in any of the following outcomes: death; a life-threatening adverse drug experience; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability/incapacity; a congenital anomaly/birth defect; an important medical event that may require medical or surgical intervention to prevent any of the above outcomes.
Time Frame: Baseline up to 46 days
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  TEAEs | 1 | 0 | 0 | 3
  SAEs | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours Post-dose (AUC0-24) of Pirtobrutinib
Description: PK: AUC0-24 of Pirtobrutinib.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24 hours post-dose)
Population: All participants who received a dose of Pirtobrutinib, had at least 1 quantifiable PK concentration of Pirtobrutinib and had at least 1 PK parameter computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL) | 84100 (27.2) | 135000 (81.8) | 200000 (22.6) | 225000 (22.3)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Hour Zero to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL) | 143000 (29.8) | 259000 (101) | 379000 (16.9) | 490000 (26.8)

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC0-inf of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL) | 144000 (30.1) | 260000 (100) | 382000 (16.9) | 492000 (26.9)

5. Secondary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Pirtobrutinib
Description: PK: %AUCextrap of pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of AUCextrap | 0.869 (39.9) | 0.504 (61.2) | 0.474 (113) | 0.458 (48.1)

6. Secondary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 6600 (28.7) | 9050 (65.9) | 13700 (32.8) | 13000 (27.1)

7. Secondary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 3.25 [1.50 to 7.00] | 2.75 [2.00 to 4.00] | 3.00 [2.50 to 7.00] | 4.01 [2.50 to 9.00]

8. Secondary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Cohort 1)
Description: PK: λZ of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib
Number analyzed (Participants) | 6
1/hour (1/h)
  Subject 1 | 0.0367
  Subject 2 | 0.0423
  Subject 3 | 0.0242
  Subject 4 | 0.0477
  Subject 5 | 0.0285
  Subject 6 | 0.0469

9. Secondary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Cohort 2)
Description: PK: λZ of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Cohort 2: 600 mg Pirtobrutinib
Number analyzed (Participants) | 6
1/hour (1/h)
  Subject 1 | 0.0322
  Subject 2 | 0.0317
  Subject 3 | 0.0381
  Subject 4 | 0.0327
  Subject 5 | 0.0353
  Subject 6 | 0.0368

10. Secondary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Cohort 3)
Description: PK: λZ of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Cohort 3: 800 mg Pirtobrutinib
Number analyzed (Participants) | 6
1/hour (1/h)
  Subject 1 | 0.0279
  Subject 2 | 0.0263
  Subject 3 | 0.0339
  Subject 4 | 0.0339
  Subject 5 | 0.0295
  Subject 6 | 0.0410

11. Secondary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Cohort 4)
Description: PK: λZ of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6
1/hour (1/h)
  Subject 1 | 0.0291
  Subject 2 | 0.0367
  Subject 3 | 0.0330
  Subject 4 | 0.0313
  Subject 5 | 0.0320
  Subject 6 | 0.0396

12. Secondary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: CL/F of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per hour (L/h) | 2.08 (30.1) | 2.31 (100) | 2.10 (16.9) | 1.83 (26.9)

13. Secondary Outcome: PK: Apparent Volume of Distribution at Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter (L) | 57.0 (23.5) | 67.1 (96.2) | 66.1 (26.4) | 54.7 (23.2)

14. Secondary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t1/2) of Pirtobrutinib
Description: PK: t1/2 of Pirtobrutinib.
Time Frame: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 19.0 (28.4) | 20.2 (7.71) | 21.9 (16.3) | 20.7 (11.2)

ADVERSE EVENTS:
Time Frame: Upto 46 days
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Cohort 1: 300 mg Pirtobrutinib | Cohort 2: 600 mg Pirtobrutinib | Cohort 3: 800 mg Pirtobrutinib | Cohort 4: 900 mg Pirtobrutinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 300 mg Pirtobrutinib (N=6) | Cohort 2: 600 mg Pirtobrutinib (N=6) | Cohort 3: 800 mg Pirtobrutinib (N=6) | Cohort 4: 900 mg Pirtobrutinib (N=6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT06181006/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT06181006/SAP_001.pdf